CLINICAL TRIAL: NCT03059173
Title: Interest of Myo-inositol Supplementation in Women With Polycystic Ovarian Syndrome During Induction of Ovulation With Clomiphene Citrate
Brief Title: Interest of Myo-inositol Supplementation in Women With Polycystic Ovarian Syndrome
Acronym: MYOPK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government); Laboratoires Besins International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015_68; 2016-A01246-45 (Other: ID-RCB number, ANSM); PHRC_N_15-0116 (Other: PHRC number)
Record Dates: First submitted 2017-01-26; First posted 2017-02-23 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Polycystic Ovary Syndrome; Reproductive Medicine
Keywords: Polycystic ovary syndrome; Reproductive medicine
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Inositol; 5-methyltetrahydrofolate; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myo-Inositol + Levomefolic acid (Experimental): The experimental group will receive the dietary supplement: 4 g of MYO + 0.736 mg of 5-MTHF, glucosamine salts per day per os (in 2 bags per day) in addition to the standard therapy (Clomiphene Citrate).
  Interventions: Dietary Supplement: Myo-Inositol + Levomefolic acid; Drug: Clomiphene Citrate
- Placebo (Placebo Comparator): The control group will receive the standard therapy ( Clomiphene Citrate) and a placebo containing only 0.736 mg of 5-MTHF, glucosamine salts
  Interventions: Drug: Clomiphene Citrate; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Myo-Inositol + Levomefolic acid — Dietary supplement Gynositol® MTHF containing myo-inositol (4 g) and Levomefolic acid on glucosamine salts(0.736 mg) in a same bags Supplementation started on average one month before treatment with Clomiphene citrate and continued throughout cycles of Clomiphene citrate (maximum 9 cycles). Treatment will be delivered during ultrasound visit at D12 of each cycle.
  Other Names: Myo + [6S]-5-MethylTetrahydrofolate(5-MTHF) ou Gynositol (R)
  Arms: Myo-Inositol + Levomefolic acid
Drug: Clomiphene Citrate — Clomiphene citrate 50 mg. taking D2 to D6 of each cycle (maximum 9 cycles). Treatment will be delivered during ultrasound visit at D12 of each cycle and the dose will be increased if necessary.
Dietary Supplement: placebo — a placebo containing only 0.736 mg of 5-MTHF, glucosamine salts
  Arms: Placebo

SUMMARY:
The main objective will be to check if MyoInositol (MYO) reduces the total resistance rate to Clomiphene Citrate (CC). For this, our study will be controlled, randomized and double blinded. It will include patients with PCOS (polycystic ovary syndrome, defined by the Rotterdam criteria) who wish to become pregnant and are eligible to simple ovulation induction by CC. Half of them will receive MYO + levomefolic acid (5-MTHF) in addition to the CC, while the other half will receive a placebo containing only 5-MTHF in addition to the CC. The MYO supplementation will be initiated at least one month before taking CC and will be continued throughout this treatment until pregnancy or before switching to another type of treatment for ovulation induction if no pregnancy is obtained after 6 ovulatory cycles.

ELIGIBILITY:
Inclusion Criteria:

* Wishing pregnancy,
* Having PCOS defined by the Rotterdam criteria: high antral follicle count (AFC) (> 19 per ovary) and/or a disorder of the cycle and/or hyperandrogenism (at least two of the three criteria),
* Having never been treated with CC (or previous treatment with CC interrupted for > 3 months).
* Having received complete information and having signed consent.
* Covered by social security

Exclusion Criteria:

* Intolerance to CC in previous treatment,
* BMI > 35,
* Other associated cause of oligoanovulation requiring specific treatment (eg., Hyperprolactinemia or functional hypothalamic anovulation),
* Ongoing pregnancy at the time of CC initiation,
* Other male or female cause of hypo-fertility,
* History of ovarian drilling,
* Negative rubella serology.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Woman of childbearing age
Enrollment: 276 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2027-09-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Total resistance rate under CC for ovulation induction in patients with PCOS. | At each cycle during 4 months
  The total resistance to CC is defined by failure to ovulate at least one time during 4 subsequent cycles in women requiring 150 mg/day from D2 to D6.

SECONDARY OUTCOMES:
Rate of responders (i.e., 100% cycles with ovulation and/or occurrence of a pregnancy) at doses of 50 and 100mg of CC | At each cycle during one year
Rate of drop out | at each cycle during one year
Cumulative incidence of clinical pregnancy (cardiac activity on ultrasound at 6 weeks of amenorrhea) | During one year
Rate of patients switched to a 2nd line treatment with exogenous gonadotropins over the whole period of the study | At each cycle during one year

CONTACTS AND LOCATIONS:
Overall Officials: Goeffrey Robin, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU de Lille hôpital Jeanne de Flandre, Lille, France

IPD SHARING:
Plan to Share IPD: No